CLINICAL TRIAL: NCT00576979
Title: Phase I-II Study of Escalating Doses of Large Field Image-Guided Intensity Modulated Radiation Therapy (IMRT) Using Helical Tomotherapy in Combination With Etoposide (VP16) and Cytoxan as a Preparative Regimen for Allogeneic Hematopoietic Stem Cell (HSC) Transplantation for Patients With Poor Risk Acute Lymphocytic Leukemia (ALL) or Poor Risk Acute Myelogenous Leukemia (AML)
Brief Title: Intensity-Modulated Radiation Therapy, Etoposide, and Cyclophosphamide Followed By Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 05021; CHNMC-05021; CDR0000579141 (Registry Identifier: NCI PDQ); NCI-2010-00427 (Registry Identifier: NCI CTRP); R01CA154491 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Level 1: 1200cGy (Experimental): 150cGy BID x Days 1-4. Total dose 1200cGy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 2: 1350cGy (Experimental): 150cGy BID Day 1-4 then 150 cGy QD Day 5. Total dose 1350cGy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 3: 1500cGy limited dose to ribs, sternum, liver, brain 1200cGy (Experimental): 150cGy BID Day 1-5. Total dose 1500Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 4: 1500cGy limited dose to liver, brain 1200cGy (Experimental): 150cGy BID Day 1-5. Total dose 1500Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 5: 1600cGy limited dose to liver, porta-hepatic, brain 1200cGy (Experimental): 160cGy BID Day 1-5. Total dose 1600Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 6: 1700cGy limited dose to liver, porta-hepatic, brain 1200cGy (Experimental): 170cGy BID Day 1-5. Total dose 1700Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 7: 1800cGy limited dose to liver, porta-hepatic, brain 1200cGy (Experimental): 180cGy BID Day 1-5. Total dose 1800Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 8: 1900cGy limited dose to liver, porta-hepatic, brain 1200cGy (Experimental): 190cGy BID Day 1-5. Total dose 1900Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy
- Level 9: 2000cGy limited dose to liver, porta-hepatic, brain 1200cGy (Experimental): 200cGy BID Day 1-5. Total dose 2000Gy.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: intensity-modulated radiation therapy; Radiation: tomotherapy

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Procedure: allogeneic bone marrow transplantation — Occurs approximately 48 hours after completion of cyclophosphamide
Procedure: allogeneic hematopoietic stem cell transplantation — Occurs approximately 48 hours after completion of cyclophosphamide
Procedure: peripheral blood stem cell transplantation — Occurs approximately 48 hours after completion of cyclophosphamide
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Radiation: tomotherapy — Undergo IMRT using helical tomotherapy
  Other Names: helical tomotherapy

SUMMARY:
RATIONALE: Giving intensity modulated radiation therapy (IMRT) and chemotherapy, such as etoposide and cyclophosphamide, before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving IMRT together with chemotherapy before transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects and best dose of intensity-modulated radiation therapy (IMRT) when given together with etoposide and cyclophosphamide followed by donor stem cell transplant and to see how well they work in treating patients with relapsed or refractory acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
OBJECTIVES: I. To establish the maximum tolerated dose [MTD] of large field image-guided IMRT, using helical tomotherapy when given in combination with intravenous cyclophosphamide and VP-16 as a preparative regimen for allogeneic hematopoietic stem cell transplantation (HSCT) from an human leukocyte antigen (HLA)-identical sibling or unrelated donor in patients with ALL or AML with induction failure or in relapse. (Phase I) II. To describe the toxicity at each dose level standard. (Phase I) III. To collect data on the radiation dose to normal organs and bone marrow using tomotherapy targeted total-body irradiation (TBI). (Phase I) IV. To estimate the overall survival probability, disease free survival probability and relapse rate associated with this regimen. (Phase II) V. To characterize the treatment related mortality and toxicity profile (early/late) associated with this regimen. (Phase II) VI. To descriptively compare the outcomes of patients treated on this protocol to a comparable patient population conditioned with whole body radiation. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of intensity-modulated radiation therapy (IMRT) followed by a phase II study.

PREPARATIVE REGIMEN: Patients undergo IMRT using helical tomotherapy once or twice daily on days -10 to -6 or -10 to -7. Patients also receive etoposide intravenously (IV) on day -6 or -5 and cyclophosphamide IV on day -4 or -3.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell or bone marrow transplantation on day -1 or day 0. After completion of study treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphocytic leukemia or acute myelogenous leukemia who are not in first or second remission (i.e., after failing remission induction therapy or in relapse or beyond second remission)
* All candidates for this study must have a human leukocyte antigen (HLA) (A, B, C, DR) identical sibling who is willing to donate bone marrow or primed blood stem cells or a 10/10 allele matched unrelated donor; a single allele mismatch at A, B, C, DR, or DQ and a KIR mismatch at C will be allowed; all ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques
* Prior therapy with VP-16, Busulfan, and Cytoxan is allowed
* A cardiac evaluation with an electrocardiogram showing no ischemic changes or abnormal rhythm and an ejection fraction of >= 50% established by multi gated acquisition scan (MUGA) or echocardiogram
* Patients must have a serum creatinine of less than or equal to 1.2 or creatinine clearance > 80 ml/min
* A bilirubin of less than or equal to 1.5
* Serum glutamic oxaloacetic transaminase (SGOT) less than 5 times the upper limit of normal
* Serum glutamate pyruvate transaminase (SGPT) less than 5 times the upper limit of normal
* Pulmonary functioning tests including diffusing capacity of carbon monoxide (DLCO) will be performed; forced expiratory volume in one second (FEV1) and DLCO should be greater than 50% of the predicted normal value
* The time from the end last induction or reinduction attempt should be >= 14 days
* Signed informed consent form approved by the Institutional Review Board (IRB) is required

DONOR: Any sibling donors who are histocompatible with the prospective recipient will be considered a suitable donor

* Donors will be excluded if for psychological or medical reasons they are unable to tolerate the procedure
* Donor should be able to donate peripheral blood stem cells or bone marrow

Exclusion Criteria:

* Prior radiation therapy that would exclude the use of total-body irradiation
* Patients who have undergone bone marrow transplantation previously and who have relapsed
* Patients with psychological or medical condition that patients physician deems unacceptable to proceed to allogeneic bone marrow transplant
* Pregnancy
* Electrocardiogram (EKG) showing ischemic changes or abnormal rhythm and/or an echocardiogram or MUGA scan showing abnormal wall motion or ejection fraction < 50%

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03-04 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2026-02-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S. Stein, MD, Study Chair — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: 1200cGy: 150cGy BID x Days 1-4. Total dose 1200cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 2: 1350cGy: 150cGy BID Day 1-4 then 150 cGy QD Day 5. Total dose 1350cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 3: 1500cGy (1200 cGy Limited Dose to Ribs, Sternum, Liver, Brain); Period 4: 1500cGy (1200 cGy Limited Dose to Liver, Brain): 150cGy BID Day 1-5. Total dose 1500Gy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 5: 1600cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain): 160cGy BID Day 1-5. Total dose 1600Gy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 6: 1700cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain): 170cGy BID Day 1-5. Total dose 1700Gy. Patient age 18-55
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 7: 1800cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain): 180cGy BID Day 1-5. Total dose 1800cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 8: 1900cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain): 190cGy BID Day 1-5. Total dose 1900cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Period 9: 2000cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain): 200 cGy BID Day 1-5. Total dose 2000cGy
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
Period: Overall Study
Arm/Group | Period 1: 1200cGy | Period 2: 1350cGy | Period 3: 1500cGy (1200 cGy Limited Dose to Ribs, Sternum, Liver, Brain) | Period 4: 1500cGy (1200 cGy Limited Dose to Liver, Brain) | Period 5: 1600cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain) | Period 6: 1700cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain) | Period 7: 1800cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain) | Period 8: 1900cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain) | Period 9: 2000cGy (1200 cGy Limited Dose to Liver, Porta-hepatic, Brain)
Started | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Level 3: 1500cGy Limited Dose to Ribs, Sternum, Liver, Brain 1200cGy; Level 4: 1500cGy Limited Dose to Liver, Brain 1200cGy: 150cGy BID Day 1-5. Total dose 1500cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Level 5: 1600cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy: 160cGy BID Day 1-5. Total dose 1600cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Level 6: 1700cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy: 170cGy BID Day 1-5. Total dose 1700cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Level 7: 1800cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy: 180cGy BID Day 1-5. Total dose 1800cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Level 8: 1900cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy: 190cGy BID Day 1-5. Total dose 1900cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Level 9: 2000cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy: 200cGy BID Day 1-5. Total dose 2000cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
- Total: Total of all reporting groups
Arm/Group | Level 1: 1200cGy | Level 2: 1350cGy | Level 3: 1500cGy Limited Dose to Ribs, Sternum, Liver, Brain 1200cGy | Level 4: 1500cGy Limited Dose to Liver, Brain 1200cGy | Level 5: 1600cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 6: 1700cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 7: 1800cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 8: 1900cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 9: 2000cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Total
Number analyzed (Participants) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 34.4 [21.6 to 44.9] | 24.5 [20.8 to 53.1] | 32.7 [22.3 to 54.8] | 31.1 [20.8 to 51.4] | 37.5 [30.1 to 53.3] | 52.5 [27.4 to 56.5] | 36.5 [19.7 to 57.7] | 38.4 [19.9 to 54.0] | 39.4 [16.5 to 50.2] | 34.4 [16.5 to 57.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 3 | 3 | 2 | 5 | 5 | 4 | 31
  Male | 2 | 2 | 2 | 3 | 3 | 4 | 1 | 1 | 2 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 10
  Black, not of Hispanic origin | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hispanic | 1 | 1 | 1 | 3 | 2 | 2 | 1 | 2 | 4 | 17
  Other, Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 1 | 5 | 3 | 2 | 3 | 4 | 1 | 2 | 22
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 51

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Intensity-modulated Radiotherapy (Phase I)
Description: Toxicities will be recorded using two distinct grading systems: the modified Bearman scale and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 3.0 scale.
Time Frame: 30 days post transplant
Measure: Number; unit: cGy
Groups:
- All Levels: 1200 cGy to 2000cGy: Patient age 18-55
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
Arm/Group | All Levels: 1200 cGy to 2000cGy
Number analyzed (Participants) | 51
cGy | 2000

ADVERSE EVENTS:
Time Frame: Up to 2 years. To be evaluable for toxicity, a patient must start treatment and be observed for at least 30 days following the completion of the transplant procedure or have experienced DLT. Hematological toxicities will be evaluated from day 0, the day the patient receives allogeneic cell transplant. No dose escalation will occur until DLT evaluations for all patients on a dose level.
Description: The modified Bearman Scale will be used to define DLT events and the CTCAE 3.0 scale will be used for reporting adverse events. CTCAE version 4.03 is used for reporting adverse events in Arm 9.
Groups:
- Level 9: 2000cGy: 200cGy BID Day 1-5. Total dose 1900cGy.
  cyclophosphamide: Given IV
  etoposide: Given IV
  allogeneic bone marrow transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  allogeneic hematopoietic stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  peripheral blood stem cell transplantation: Occurs approximately 48 hours after completion of cyclophosphamide
  intensity-modulated radiation therapy: Undergo IMRT
  tomotherapy: Undergo IMRT using helical tomotherapy
Arm/Group | Level 1: 1200cGy | Level 2: 1350cGy | Level 3: 1500cGy Limited Dose to Ribs, Sternum, Liver, Brain 1200cGy | Level 4: 1500cGy Limited Dose to Liver, Brain 1200cGy | Level 5: 1600cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 6: 1700cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 7: 1800cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 8: 1900cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy | Level 9: 2000cGy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/9 | 3/6 | 0/6 | 0/6 | 1/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 9/9 | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: 1200cGy (N=3) | Level 2: 1350cGy (N=3) | Level 3: 1500cGy Limited Dose to Ribs, Sternum, Liver, Brain 1200cGy (N=9) | Level 4: 1500cGy Limited Dose to Liver, Brain 1200cGy (N=6) | Level 5: 1600cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 6: 1700cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 7: 1800cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 8: 1900cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 9: 2000cGy (N=6)
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
10040047-Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10005364-Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Toxicity (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
10038695-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10065746-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: 1200cGy (N=3) | Level 2: 1350cGy (N=3) | Level 3: 1500cGy Limited Dose to Ribs, Sternum, Liver, Brain 1200cGy (N=9) | Level 4: 1500cGy Limited Dose to Liver, Brain 1200cGy (N=6) | Level 5: 1600cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 6: 1700cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 7: 1800cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 8: 1900cGy Limited Dose to Liver, Porta-hepatic, Brain 1200cGy (N=6) | Level 9: 2000cGy (N=6)
10002272-Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Edema:head and neck (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4 | 3 | 0 | 3 | 4 | 0
Edema:limb (Blood and lymphatic system disorders) | 2 | 1 | 7 | 6 | 6 | 5 | 6 | 6 | 0
Edema:trunk/genital (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 | 2 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphatics - Other (Specify, __) LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 9 | 6 | 6 | 3 | 0 | 5 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 2 | 9 | 5 | 6 | 5 | 6 | 6 | 0
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelets (Blood and lymphatic system disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
10040741-Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10040752-Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Cardiac Arrhythmia - Other (Specify, __) TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cardiac Toxicity (Cardiac disorders) | 0 | 1 | 3 | 3 | 1 | 1 | 2 | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0 | 4 | 4 | 1 | 2 | 3 | 3 | 0
Hypotension (Cardiac disorders) | 1 | 2 | 6 | 5 | 2 | 4 | 3 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 | 1 | 7 | 6 | 3 | 1 | 6 | 6 | 0
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
10005886-Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye syndrome (Eye disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 0
Ocular/Visual - Other (Specify, __) CLOUDINESS LEFT CORNEA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular/Visual - Other (Specify, __) EYES STAY OPEN (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular/Visual - Other (Specify, __) PALLOR OF CONJUNCTIVAE (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular/Visual - Other (Specify, __) SCLERAL ICTERUS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision-blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Watery eye (epiphora, tearing) (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
10000081-Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10003445-Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10009887-Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10010774-Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10012727-Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10013781-Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10013946-Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10013950-Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10017853-Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10028130-Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10028813-Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10031009-Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10047700-Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10051746-Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10065721-Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 2 | 3 | 9 | 6 | 6 | 6 | 5 | 5 | 0
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 0 | 2 | 4 | 2 | 0
Dehydration (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 8 | 6 | 6 | 6 | 6 | 6 | 0
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 | 0 | 5 | 3 | 4 | 1 | 1 | 2 | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 2 | 2 | 3 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 0
Gastrointestinal - Other (Specify, __) BELCHING (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) CHANGE IN BOWEL HABITS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) FREQUENT BOWEL MVMT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal - Other (Specify, __) GI UPSET (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) LICHENOID CHANGES IN MOUTH (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) MOUTH SORE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) PERIANAL NUMBNESS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GI Toxicity (Gastrointestinal disorders) | 2 | 3 | 6 | 3 | 6 | 2 | 6 | 5 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 5 | 2 | 2 | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Incontinence, anal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 | 3 | 9 | 5 | 5 | 4 | 5 | 6 | 0
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2 | 1 | 9 | 5 | 4 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 9 | 4 | 6 | 6 | 6 | 6 | 0
10008531-Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10014222-Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10016059-Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10016256-Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10016558-Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
10017577-Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10018065-General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10033371-Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10050068-Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10051792-Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10062501-Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 | 3 | 8 | 6 | 6 | 6 | 6 | 6 | 0
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 | 2 | 6 | 3 | 3 | 3 | 3 | 4 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (General disorders) | 0 | 1 | 7 | 3 | 4 | 5 | 6 | 4 | 0
Pain (General disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Pain - Other (Specify, __) GENERALIZED BODYACHE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (Specify, __) GENERALIZED PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (Specify, __) JAW PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain - Other (Specify, __) L/R SIDE BODY PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain - Other (Specify, __) MANDIBULAR (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (Specify, __) PICC LINE SITE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (Specify, __) PICC SITE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (Specify, __) TOOTH (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain CHEST NOS LEFT SIDE (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rigors/chills (General disorders) | 2 | 2 | 7 | 5 | 2 | 4 | 3 | 5 | 0
Syndromes - Other (Specify, __) ENGRAFTMENT SYN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syndromes - Other (Specify, __) ENGRAFTMENT SYNDROME (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight gain (General disorders) | 2 | 0 | 3 | 3 | 1 | 0 | 1 | 0 | 0
Weight loss (General disorders) | 1 | 1 | 7 | 3 | 4 | 2 | 2 | 2 | 0
Hepatic Toxicity (Hepatobiliary disorders) | 0 | 1 | 3 | 2 | 2 | 0 | 0 | 1 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
10021881-Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10040753-Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10046914-Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10058838-Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10061229-Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Febrile neutropenia (Infections and infestations) | 1 | 1 | 4 | 2 | 0 | 1 | 0 | 0 | 0 — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection - Other (Specify, __) CMV INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 2 | 7 | 3 | 3 | 3 | 0 | 3 | 0 — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 0
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Stomatitis (Infections and infestations) | 2 | 1 | 8 | 5 | 4 | 0 | 0 | 4 | 0
10006504-Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10061103-Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10000636-Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10001551-Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
10001675-Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10003481-Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10005364-Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10011368-Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10022402-INR increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10025256-Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10029366-Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10035528-Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10047896-Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10047900-Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10049182-White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10055599-Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10056910-GGT increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10059895-Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10000486-Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10001680-Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10002646-Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10020680-Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10021018-Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10021038-Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 | 3 | 6 | 5 | 4 | 3 | 6 | 4 | 0
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 | 3 | 7 | 5 | 6 | 6 | 5 | 6 | 0
Amylase (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 | 3 | 7 | 6 | 6 | 5 | 6 | 5 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 | 2 | 8 | 6 | 5 | 4 | 5 | 6 | 0
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 2 | 2 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 2 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 5 | 6 | 0
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2 | 3 | 1 | 2 | 0 | 0
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Creatinine (Metabolism and nutrition disorders) | 0 | 2 | 5 | 2 | 1 | 4 | 5 | 3 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 | 3 | 8 | 6 | 6 | 4 | 0 | 5 | 0
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 0
Lipase (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 1 | 2 | 1 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Metabolic/Laboratory - Other (Specify, __) CARBON DIOXIDE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic/Laboratory - Other (Specify, __) HYPOVITAMINOSIS D (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Metabolic/Laboratory - Other (Specify, __) HYPOGAMMAGLOBINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic/Laboratory - Other (Specify, __) HYPOGAMMAGLOBULINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 | 2 | 8 | 6 | 5 | 2 | 4 | 6 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 0 | 1 | 3 | 4 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Proteinuria (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 0
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 | 3 | 8 | 5 | 6 | 6 | 6 | 6 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 2 | 2 | 2 | 2 | 0
10029104-Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10013573-Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10013911-Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10019211-Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10020765-Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10027175-Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10029205-Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10033987-Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10041349-Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10044565-Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Apnea (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 3 | 2 | 1 | 2 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurology - Other (Specify, __) DISORIENTED (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurology - Other (Specify, __) LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurology - Other (Specify, __) NUMBNESS (B) FEET (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurology - Other (Specify, __) PERIPHERAL NEUROP. (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurology - Other (Specify, __) RIGHT FACIAL NUMBNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy: sensory (Nervous system disorders) | 2 | 0 | 5 | 3 | 2 | 2 | 1 | 1 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Syncope (fainting) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 2 | 3 | 0 | 3 | 0 | 5 | 0
10001497-Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10002855-Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10010300-Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10012260-Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10012378-Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10019077-Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10022437-Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10037175-Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10038743-Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (children <3 years of age) (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Mood alteration (Psychiatric disorders) | 3 | 3 | 8 | 5 | 4 | 4 | 4 | 5 | 0
Neurology - Other (Specify, __) ALTERED MENTAL STATUS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
10046539-Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10069339-Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder Toxicity (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal Toxicity (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Renal/Genitourinary - Other (Specify, __) DYSURIA (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal/Genitourinary - Other (Specify, __) MILD RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Urine color change (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
10046901-Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10046916-Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10061339-Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sexual/Reproductive Function - Other (Specify, __) VAGINAL ITCHING (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10020201-Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10038695-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
10065746-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 7 | 3 | 3 | 4 | 3 | 3 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3 | 3 | 3 | 2 | 0
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) CHEST CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) NASAL DISCHARGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) TACHPNEIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) TACHYPNEIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) WEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10015277-Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10033474-Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10037847-Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
10040865-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
10040868-Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
10054524-Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Dermatology/Skin - Other (Specify, __) ABRASION-LOWER THIGHS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Specify, __) BUMPS - BUTTOCK AREA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) CONTUSION - HEAD (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) DARKNESS OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) FOLLICULITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Specify, __) ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) PALE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) PALLOR OF FACE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) PEELING OF FINGERS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) PEELING OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) SCALP LESIONS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Specify, __) SEBORRHEIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Specify, __) SKIN ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatology/Skin - Other (Specify, __) SKIN PEELING (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Specify, __) SKIN SENSITIVITY (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) SKIN TEAR RLQ (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 7 | 3 | 3 | 5 | 2 | 3 | 0
Flushing (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 6 | 4 | 1 | 4 | 0 | 0
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 4 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 5 | 6 | 6 | 5 | 4 | 5 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 | 2 | 6 | 2 | 3 | 1 | 0 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 5 | 3 | 6 | 4 | 6 | 0
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 2 | 7 | 6 | 6 | 6 | 6 | 5 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 — Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 0
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
10020772-Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
10021097-Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemorrhage, GI (Vascular disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 3 | 0 | 0
Hemorrhage, GU (Vascular disorders) | 0 | 2 | 6 | 4 | 3 | 0 | 3 | 2 | 0
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 1 | 0 | 4 | 1 | 2 | 3 | 2 | 0 | 0
Hemorrhage/Bleeding - Other (Specify, __) RETINAL HEMORRHAGE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhage/Bleeding - Other (Specify, __) RIGHT EYE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhage/Bleeding - Other (Specify, __) RIGHT RETINAL HEMORRHAGE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
PTT (Partial Thromboplastin Time) (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic microangiopathy (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No